CLINICAL TRIAL: NCT04415957
Title: Elastic Tape Reduces Dyspnea and Improves Health Status, and Health-related Quality of Life in Non-obese COPD Males: a Randomized Controlled Trial
Brief Title: Elastic Tape Relieves Symptoms and Improves Health-related Quality of Life in COPD (Chronic Obstructive Pulmonary Disease)
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETPADCOPD
Record Dates: First submitted 2020-02-17; First posted 2020-06-04 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; dyspnea; respiratory mechanics; exercise capacity; physical activity; elastic tape
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization sequence was computer-generated and implemented by an investigator not involved in recruitment, assessment, or treatment. Concealment allocation was assured by placing the randomization in opaque envelopes sequentially numbered. An envelope for every participant was opened in sequential order after baseline assessments. The participants and physical therapists who performed the intervention could not be blinded due to the nature of the intervention. However, all the outcomes and statistical assessors were blinded to group allocation and previous test results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Tape Group (ETG) (Experimental): The ET placement was previously described by Pinto et al. (2020). Briefly, the subject's trunk was passively extended for ET placement. The ET was placed considering the origins and insertions of the following muscles: rectus abdominis, internal oblique, and internal intercostal. ET has shown six days of durability on average, so the participants were asked to return to change the ET after seven days.
  Interventions: Other: Elastic Tape
- Control Group (CG) (No Intervention): CG received instructions about the importance of becoming physical activity. Furthermore, the participants included in CG were invited to place the ETs at the end of the protocol.

INTERVENTIONS:
Other: Elastic Tape — The subject's trunk was passively extended for ET placement. The ET was placed on the chest wall and abdomen, considering the origins and insertions of the following muscles: rectus abdominis, internal oblique, and internal intercostal. The intervention lasted 14 days, therefore, the participants remained with the tapes for two consecutive weeks. Due to the adhesive durability of ETs (6 weeks on average), the participants were asked to return to change the ET after seven days.
  Arms: Elastic Tape Group (ETG)

SUMMARY:
* The goal of this randomized controlled trial is to investigate the effects of elastic tape in individuals with mild to very severe COPD.
* The main questions it aims to answer are:

Does the ET influence on daily life physical activity (DLPA), dyspnea, health status, health-related quality of life (HRQoL), and anxiety and depression symptoms in individuals with COPD?

Does the ET modify the perceived barriers to DLPA in individuals with COPD?

* The protocol lasted 21 days, including seven days of initial assessments and 14 days of intervention. Before baseline assessments, participants were randomly allocated into intervention (Elastic Tape Group, ETG, n=25) or control groups (CG, n=25). The ETG received ETs on the chest wall and abdomen for two consecutive weeks while the CG received instructions about the importance of becoming physical activity. The assessments were performed before and after 14 days of intervention.
* The ET placement was previously described by Pinto et al. (2020).

DETAILED DESCRIPTION:
Background: The elastic tape (ET) is a novel intervention that has been shown to improve exercise capacity acutely in laboratory tests; however, its effect on a patient's daily life remains poorly known.

Research Question: Does the ET influence on daily life physical activity (DLPA), dyspnea, health status, and health-related quality of life (HRQoL) in individuals with COPD?

Study Design and Methods: Fifty non-obese males with moderate to very severe COPD were randomly allocated to intervention (ETG) or control groups (CG). Eligible individuals were invited to participate after a regular medical visit and randomized into two groups. The protocol lasted 21 days, including seven days of initial assessments and 14 days of intervention. The ETG received the ET positioned in the chest wall and abdomen for 14 days while CG received the usual care. Dyspnea symptoms (Transition dyspnea index, TDI; and modified Medical Research Council, mMRC) were evaluated at baseline (day 0 of protocol, visit 1), day 7 of protocol (visit 2) and day 14 of protocol (visit 3). DLPA (accelerometry), health status (COPD assessment test, CAT), and HRQoL (CRQ) were evaluated before and after the intervention. All outcomes were reassessed after seven days (day 14 of protocol, visit 3). CG received instructions about the importance of becoming physical activity. In addition, CG also had 3 visits and performed the same assessments as the ETG. At the end of protocol, the participants of CG were invited to place the ETs.

Sample size and data analysis: The sample size was calculated from a pilot study. The primary outcome used was the number of step-counts (2,800±3,500, mean (MD) ± standard deviation (SD)). A sample size of 25 participants per group was obtained to detect between-group differences (α=0.05, 1-β=0.8). Group and time interactions were assessed using a two-way repeated-measures analysis of variance (ANOVA) followed by a post hoc test of Holm-Sidak. Non-parametric data were tested by the corresponding non-parametric tests. Data were analyzed according to the intention-to-treat principle, and missing values were imputed by the expected maximization (EM) technique, using IBM SPSS Statistics for Windows (version 22). Altogether, two participants who lost follow-up had their data imputed, and one patient that exacerbated during the study was reassessed after discharge.

Results: No between-group differences were observed at baseline. ET reduced the dyspnea symptoms in all TDI domains (functional, task, and effort) and on the mMRC after 14 days compared with CG, reaching a minimal clinically important difference (≥1.0, MCID). In addition, patients in the ETG improved their CAT score compared to the CG, reaching MCID (≤2). The ETG also improved by reaching MCID in most CRQ domains (total, fatigue, emotional, and mastery) on day 14. No differences were observed in DLPA.

Conclusion: ET reduces dyspnea and improves the health status and quality of life in non-obese males with moderate to very severe COPD at mid-term. This novel and low-cost intervention can improve COPD symptoms in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Mild to severe COPD diagnosis (according to the GOLD 2022 classification);
* Males;
* Non-obese (BMI≤29.9kg/m2);
* Former smokers;
* Clinically stable (i.e.,without exacerbations for at least 30 days);
* In medical follow-up at a University tertiary hospital specialized for COPD assistance
* Consent to participate voluntarily in the study and signed the Patients' consent form.

Exclusion Criteria:

* Asthma-COPD overlap;
* Continuous use of oxygen therapy;
* Postoperative thoracic surgery;
* Open wounds or skin diseases on the chest or abdomen;
* Allergic skin reactions to the use of adhesive bandages, plasters, or other adhesive materials;
* Cardiovascular or musculoskeletal disease that compromise any assessments;
* Undergoing pulmonary rehabilitation(PR);
* Participating in other research studies;
* Unability to understand our questionnaire.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change in daily life physical activity (DLPA) | Change from baseline physical activity levels after 14 days of intervention
  Participants were instructed to wear the device for the waking hours of seven consecutive days, removing it only during swimming activities. A valid DLPA day was considered when the device had at least eight hours of data collection. In addition, every individual had at least five days per week. DLPA and sedentary time intensity were classified by the total activity counts accumulated in 60-s epoch length with the normal signal processing filter and sampling frequency of 60Hz. The Troiano et al. (2008) algorithm cut points were applied to set DLPA. Data were presented as the average number of steps per day (steps/day), time spent in moderate to vigorous physical activities (MVPA, minutes/day), and sedentary time, expressed as the percentage of waking hours.

SECONDARY OUTCOMES:
Change in dyspnea | Change from baseline dyspnea at 7th and 14th days of intervention
  Two different dyspnea scales were used modified Medical Research Council (mMRC) and Baseline and Transitional dyspnea index (BDI/TDI).
  The mMRC is a unidirectional 0-4-point scale whose questions closely match daily activities that provoke dyspnea. It has also been used in clinical practice to categorize COPD symptomatic burden and provide useful information about COPD-induced disability.
  The BDI/TDI questionnaire is a multidimensional assessment of dyspnea. The BDI/TDI has been widely validated in COPD and remains the most frequently used questionnaire in clinical research, particularly for therapeutic trials. BDI/TDI evaluates dyspnea in three domains: functional impairment, the magnitude of the task, and the magnitude of effort. The change of 1.0 point is considered a minimal clinically important difference (MCID). The higher the score in TDI, the greater the improvement in dyspnea.
Change in health status | Change in health status after 14 days of intervention
  Health status was assessed using the COPD Assessment Test (CAT). CAT aims to measure the impact of COPD on a patient's health status. The items include physical symptoms (cough, phlegm, chest tightness, breathlessness), activity limitation, energy besides confidence in leaving home, and sleep quality. CAT has a total maximum score of 40 points (maximum impairment). Scores from 0 to 10, 11 to 20, 21 to 30, and 31 to 40 represent mild, moderate, severe, or very severe clinical impact, respectively. A change of -2.54 points is considered a MCID.
Change in health-related quality of life (HRQoL) | Change in HRQoL after 14 days of intervention
  HRQoL was assessed using the Chronic Respiratory Questionnaire (CRQ). The CRQ is a validated questionnaire developed to evaluate the effects of treatments on quality of life in clinical trials and has been validated in Brazilian-Portuguese. The CRQ comprises four domains: dyspnea, fatigue, emotional function, and mastery. An MCID has been determined as 0.5 for each mean domain score, and higher scores indicate improvement in HRQoL.
Change in anxiety and depression symptoms | Change from baseline anxiety and depression symptoms after 14 days of intervention
  The anxiety and depression symptoms were assessed by the Hospital Anxiety and Depression scale (HADs), which consists of 14 items divided into two subscales (seven questions for anxiety and seven for depression). Each item is scored from 0 to 3, with a maximum score of 21 points for each subscale. A score greater than 9 in each subscale suggests a probable clinical diagnosis of either anxiety and/or depression.
Change in barriers to daily life physical activity (DLPA) | Change in barriers to DLPA after 14 days of intervention
  The barriers to physical activity were evaluated by a questionnaire developed by Amorim et al.(2014) for patients with COPD. The questionnaire consists of 21 items rated from 0 to 3 (0= never; 3= always) divided into seven domains: lack of time, social influence, lack of energy, lack of will, fear of injury, lack of skill, and lack of structure. The score per domain ranges from 0 to 9, with a maximum of 63 points. Higher scores indicate a greater barrier, and scores greater than five are considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Celso RF Carvalho, PhD, Study Director — University of São Paulo General Hospital
Locations (1):
- Clinical Hospital of São Paulo University medical school (HCFMUSP), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pinto TF, Fagundes Xavier R, Lunardi AC, Marques da Silva CCB, Moriya HT, Lima Vitorasso R, Torsani V, Amato MBP, Stelmach R, Salge JM, Carvalho-Pinto RM, Carvalho CRF. Effects of elastic tape on thoracoabdominal mechanics, dyspnea, exercise capacity, and physical activity level in nonobese male subjects with COPD. J Appl Physiol (1985). 2020 Sep 1;129(3):492-499. doi: 10.1152/japplphysiol.00690.2019. Epub 2020 Jul 23. PMID 32702276
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] von Leupoldt A, Reijnders T, Schuler M, Wittmann M, Jelusic D, Schultz K. Validity of a Self-administered Questionnaire Version of the Transition Dyspnea Index in Patients with COPD. COPD. 2017 Feb;14(1):66-71. doi: 10.1080/15412555.2016.1246522. Epub 2016 Nov 14. PMID 27841688
- [Background] Mahler DA, O'Donnell DE. Recent advances in dyspnea. Chest. 2015 Jan;147(1):232-241. doi: 10.1378/chest.14-0800. PMID 25560861
- [Background] Dodd JW, Hogg L, Nolan J, Jefford H, Grant A, Lord VM, Falzon C, Garrod R, Lee C, Polkey MI, Jones PW, Man WD, Hopkinson NS. The COPD assessment test (CAT): response to pulmonary rehabilitation. A multicentre, prospective study. Thorax. 2011 May;66(5):425-9. doi: 10.1136/thx.2010.156372. Epub 2011 Mar 12. PMID 21398686
- [Background] Smid DE, Franssen FM, Houben-Wilke S, Vanfleteren LE, Janssen DJ, Wouters EF, Spruit MA. Responsiveness and MCID Estimates for CAT, CCQ, and HADS in Patients With COPD Undergoing Pulmonary Rehabilitation: A Prospective Analysis. J Am Med Dir Assoc. 2017 Jan;18(1):53-58. doi: 10.1016/j.jamda.2016.08.002. Epub 2016 Sep 10. PMID 27624705
- [Background] Williams JE, Singh SJ, Sewell L, Guyatt GH, Morgan MD. Development of a self-reported Chronic Respiratory Questionnaire (CRQ-SR). Thorax. 2001 Dec;56(12):954-9. doi: 10.1136/thorax.56.12.954. PMID 11713359
- [Background] Moreira GL, Pitta F, Ramos D, Nascimento CS, Barzon D, Kovelis D, Colange AL, Brunetto AF, Ramos EM. Portuguese-language version of the Chronic Respiratory Questionnaire: a validity and reproducibility study. J Bras Pneumol. 2009 Aug;35(8):737-44. doi: 10.1590/s1806-37132009000800004. PMID 19750325
- [Background] Cullen K, Talbot D, Gillmor J, McGrath C, O'Donnell R, Baily-Scanlan M, Broderick J. Effect of Baseline Anxiety and Depression Symptoms on Selected Outcomes Following Pulmonary Rehabilitation. J Cardiopulm Rehabil Prev. 2017 Jul;37(4):279-282. doi: 10.1097/HCR.0000000000000258. PMID 28640172
- [Background] Amorim PB, Stelmach R, Carvalho CR, Fernandes FL, Carvalho-Pinto RM, Cukier A. Barriers associated with reduced physical activity in COPD patients. J Bras Pneumol. 2014 Oct;40(5):504-12. doi: 10.1590/s1806-37132014000500006. PMID 25410838